CLINICAL TRIAL: NCT05740579
Title: The Danish TURNER Cryopreservation Study
Acronym: DANTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DANTEcryo
Record Dates: First submitted 2022-12-14; First posted 2023-02-23 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Fertility Disorders; Turner Syndrome; Premature Ovarian Failure
MeSH Terms: conditions — Turner Syndrome; Primary Ovarian Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: laparoscopic cryopreservation of one ovary — Laparoscopic removal of one ovary as child. In adulthood cortical tissue is replaced in the abdomen in order to improve fertility and pregnancy rates in Turner syndrome women.

SUMMARY:
The goal of this clinical trial is to investigate if cryopreservation of ovarian tissue in girls with Turner syndrome can improve their fertility and lead to increased number of liveborn babies of Turner syndrome mothers. Women with Turner syndrome suffer from premature ovarian insufficiency which leads to infertility and lack of estrogen.

The main questions it aims to answer are:

* Does the number of pregnancies and liveborn children increase after cryopreservation of ovarian tissue in turner syndrome?
* Is the possible to predict when a girl with Turner syndrome reach menopause using monitoring of sex hormones?
* Is it possible to identify any genes causing ovarian failure in Turner syndrome females?

Participants between 2-18 years old will be asked to participate in a laparoscopic surgery and removal of one ovary in order to cryopreserve the tissue until adulthood. The the cortical tissue will be autotransplanted in order to preserve fertility. The participant will during the study period be monitored using sex hormones.

Furthermore, the investigators wish to investigate the ovarian tissue using RNA sequencing and DNA methylation analysis.

No comparison group is present.

DETAILED DESCRIPTION:
Hypothesis:

The majority of patients with Turner Syndrome (TS) lose their ovarian germ cells early in life. The primary hypothesis is that some patients with TS can become pregnant with their own oocytes after undergoing cryopreservation of one ovary during childhood, followed by auto-transplantation in adulthood.

Introduction Hypergonadotropic hypogonadism is a consistent trait in Turner syndrome (TS) affecting up to 95%. Through decades, a TS diagnosis was equivalent to a life with infertility. Despite a broad range of several other comorbidities, dealing with infertility is one of the most detrimental factors affecting quality of life in TS.

Most girls and women with TS undergo premature ovarian failure or insufficiency (POI) during childhood or early adolescence, before sufficient pubertal maturation. Spontaneous menarche is only present in 4-12% of 45,X females, although more frequent among mosaic karyotypes. Only a minority continue to have regular menstrual cycles (3-9%, depending on karyotype).

According to international guidelines, TS girls should be treated with estrogen from the age of 11-12 years old and later progesterone is added to ensure breakthrough bleedings. Besides ensuring uterine growth, estrogen has a wide range of beneficial effects across the entire body and receptors are present in most tissues. Estrogen therapy is essential in order to obtain optimal uterine growth and endometrial development ideal for embryo transfer during adult life.

During normal development of the female foetus, formation of germ cells and oocytes begins shortly after sexual differentiation at gestational week 6, reaching a maximum of up to five million germ cells by week 8-12. In second trimester, germ cells of the human ovary enter meiosis. This marks the end of formation of additional oocytes. During second and third trimester of the normal pregnancy a gradual loss of oocytes occurs, being reduced to approximately 400.000 oocytes at birth. In TS, the tipping point of germ cell creation and depletion seems to occur at the same time as in eukaryotic women, however, presumably at a much more accelerated speed. Both oogenesis and in particular folliculogenesis is compromised in TS females. In ovaries from 45,X TS foetuses, oogonia were observed, however with no occurrence of primordial, preantral, or antral follicles compared with eukaryotic female foetal ovaries, and connective tissue predominates in the ovaries. Some TS foetuses might even reach depletion before or around birth. Nevertheless, the majority probably reaches "menopause" during childhood or early adulthood. In postnatal ovaries, the presence of follicles is related to karyotype, age, signs of spontaneous puberty, and serum concentrations of gonadotropins and anti-Müllerian hormone (AMH), with 26%-60% of ovaries presenting with some follicles histologically in girls and young women with TS. In one study a high rate of abnormal follicle morphology was seen, and follicle fluid from small antral follicles had lower concentrations of estrogen and testosterone and higher concentrations of AMH compared with controls.

Peek et al investigated 46 oocytes in 10 TS women discovering that most oocytes were eukaryotic (90%), while the granoulosa cells were largely monosomic, demonstrating mosaicism confined to within the ovaries. This reveals that the ovarian content of X chromosome material is not always equivalent to the karyotypes performed on lymphocytes from a blood sample.

The take home message being that the karyotype is not always associated with oocyte quantity. Thus, follicles from 45,X women may be available and useable for assisted reproductive techniques. X chromosome monosomy and infertility is undoubtedly intertwined, and X chromosome deletions and X-autosome balanced translocations have been associated with POI, thus giving rise to the definition of a POI critical region from Xq13-Xq21 (POI2) to Xq23-q27 (POI1). Several candidate genes on the X chromosome have been suggested to contribute to ovarian function in Turner syndrome. In particular KDM6A, USP9X, ZFX, BMP15. KDM6A (a histone demethylase) is involved in gonadal dysgenesis, reestablishment of pluripotency and germ cell development. The gene is both differentially expressed and methylated in Turner syndrome.

Haploinsufficiency is associated with altered histone modifications potentially affecting transcriptional regulation of genes central for reproduction. USP9X escapes X inactivation and is a ubiquitin specific protease. Disturbances of ubiquitin are considered a plausible mechanism for disturbed oogenesis because the Drosophila orthologue of USP9X is required for eye development and oogenesis. USP9X is differentially methylated in Turner syndrome. ZFX is a DNA binding gene, which acts as a transcriptional factor. Knockout of ZFX in mice is related to decreased number of germ cells in both males and females (29). ZFX is differentially expressed in TS compared with control females (27, 30). BMP15 encodes bone morphogenetic protein 15, which stimulates AMH synthesis and folliculogenesis and is expressed in the oocyte. It belongs to a large family of proteins that play a regulating role in ovarian function. BMP15 knockout female mice are subfertile with decreased ovulation rates (32). Lastly, it has been proposed that epigenetic modifications in itself lead to ovarian failure. Hence that XIST, through X inactivation, plays a pivotal role in regulation of ovarian functioning by the X chromosome. However, most analyses to date are performed on blood from TS adults. Gene expression from TS ovarian tissue has still to be investigated to establish a reliable evidence for the pathophysiology of infertility in TS.

Fertility predictors in TS:

The question remains how to predict which TS women may be eligible for fertility treatment using own oocytes and which should immediately be referred to other options such as adoption or oocyte donation. In eukaryotic females, AMH and antral follicle count, assessed by vaginal ultrasound, are used as predictive markers of fertility.

Measurement of AMH has also been applied to TS women and correlates significantly with ovarian function in pubertal TS girls (12- 25 years). AMH levels are associated with karyotype, spontaneous pubertal development, LH/FSH values and the presence of follicles. Hence it seems useful as a tool for assessing the ovarian reserve in pubertal TS girls. However, in one study performing oocyte cryopreservation in seven TS women, there was no correlation between antral follicle count, AMH or oocytes retrieved. Oocytes were available in all seven TS girls despite low AMH concentrations.

So far, no evidence exists towards the use of AMH in younger pre-pubertal girls, and since the ovarian demise starts at an early age, there is a need for a predictive marker of future fertility in younger TS children. Since inhibin B is secreted from the developing follicles during mid-childhood, it has been suggested as a predictor of ovarian function in prepubertal children with Turner syndrome. It is believed that serum AMH and inhibin B levels reflect ovarian reserve independent from the hypothalamic-pituitary gonadal axis. Spontaneous puberty has been correlated with higher levels of AMH and inhibin B. However, inhibin B has been detectable without any signs of spontaneous puberty in TS women.

Assisted reproductive techniques:

Oocyte cryopreservation is not preferred in women with Turner syndrome, since it is only applicable during a short time-window from post-puberty until ovarian decline. The procedure requires ovarian stimulation therapy, trans-vaginal ultrasound scans as well as retrieval of a limited number of oocytes. Hence, this method can only be applied in a very small subgroup of TS women. In contrast, ovarian tissue cryopreservation (OTC) seems promising to retain fertility in TS women. The big advantage being that it can be applied to a larger age group (from 2 years and up) and independent of pubertal stage. The disadvantage being, that it requires a surgical procedure performed in preferable young children. OTC has led to live-born children in surviving cancer patients. However, in TS the procedure is still experimental. So far, OTC in TS women has been performed in a small cohort from Denmark, Canada, the Netherlands, and Sweden, but this is not yet a clinical standard procedure, but internationally cryopreservation protocols are recommended.

ELIGIBILITY:
Inclusion Criteria:

* 45,X karyotype or other Turner variant karyotypes (45,X/46,XX mosaicism, ring X mosaicism, isochromosome X)
* Age 2-17 years old
* Ability to participate in a physical examination including a cardiac examination.
* Signed consent from both parents.

Exclusion Criteria:

* Severe cardiac disease which inhibits safe surgery and pregnancy.
* Karyotype with Y chromosome material
* Mental retardation

Ages: 2 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2051-01-01 (Estimated); Study Completion 2051-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of pregnancies in Turner syndrome women | 20 to 30 years after cryopreservation
  The number of pregnancies
Number of miscarriages in pregnant Turner syndrome women | 20 to 30 years after cryopreservation
  The number of miscarriages
Number of liveborn children birthed by Turner syndrome women | 20 to 30 years after cryopreservation
  The number of liveborn children

SECONDARY OUTCOMES:
Number of ovarian follicles. | 2-5 days after surgery
  The number of primordial follicles/mm3 in ovarian tissue.
To evaluate predictors of premature ovarian failure in Turner syndrome under 18 years after ovarian cryopreservation. | From the date of inclusion in study until autotransplantation. Timeframe can be up to 30 years
  blood concentration of FSH meassured from a yearly blood sample.
To evaluate predictors of premature ovarian failure in Turner syndrome under 18 years after ovarian cryopreservation. | From the date of inclusion in study until autotransplantation. Timeframe can be up to 30 years
  Blood concentration of LH meassured from a yearly blood sample.
To evaluate predictors of premature ovarian failure in Turner syndrome under 18 years after ovarian cryopreservation. | From the date of inclusion in study until autotransplantation. Timeframe can be up to 30 years
  blood concentration of AMH meassured from a yearly blood sample.
To evaluate predictors of premature ovarian failure in Turner syndrome under 18 years after ovarian cryopreservation. | From the date of inclusion in study until autotransplantation. Timeframe can be up to 30 years
  blood concentration of Inhibin B meassured from a yearly blood sample.
To evaluate predictors of premature ovarian failure in Turner syndrome under 18 years after ovarian cryopreservation. | From the date of inclusion in study until autotransplantation. Timeframe can be up to 30 years
  blood concentration of estradiol meassured from a yearly blood sample.
To evaluate predictors of premature ovarian failure in Turner syndrome under 18 years after ovarian cryopreservation. | From the date of inclusion in study until autotransplantation. Timeframe can be up to 30 years
  blood concentration of androstenedione meassured from a yearly blood sample.
DNA Methylation in leukocytes before and after menopause | From the date of inclusion in study until autotransplantation. Timeframe can be up to 35 years.
  DNA is extracted
DNA methylation, RNA expression and proteome profile in oocytes. | At ovarian cryopreservation. Timeframe can be 1 to 15 years, an average of 3 years.
  To examine global DNA methylation, RNA expression and proteome profile in oocytes, granulosa and theca cells using single cell sequencing and spatial transcriptomics
TGF-β signaling in follicular fluid | At ovarian cryopreservation. Timeframe can be 1 to 15 years, an average of 3 years.
  To examine TGFβ signaling and steroidogenesis in theca cells, granulosa cells and follicular fluid from small antral follicles.
Maturation of follicles in vitro. | At ovarian cryopreservation. Timeframe can be 1 to 15 years, an average of 3 years.
  To investigate the ability of small antral follicles from TS patients to mature in vitro.
Evaluation of uterine growth after OTC. | From the date of inclusion in study until fertility treatment/pregnancy. Timeframe can be up to 35 years.
  By MRI
To examine somatic mosaicism in epithelial cells in the mouth. | At ovarian cryopreservation. Timeframe can be 1 to 15 years, an average of 3 years.
  FISH karyotyping of tissue from buccal swabs
To examine somatic mosaicism in peripheral lymphocytes | At ovarian cryopreservation. Timeframe can be 1 to 15 years, an average of 3 years.
  FISH karyotyping of lymphocytes from blood sample
To examine somatic mosaicism in germ cells. | At ovarian cryopreservation. Timeframe can be 1 to 15 years, an average of 3 years.
  FISH karyotyping of germ cells from ovarian biopsies.
To examine occurrence of surgical complications after OTC. | At ovarian cryopreservation. Timeframe can be 1 to 15 years, an average of 3 years.
  The number of infected Turner syndrome females after cryopreservation
To examine occurrence of surgical complications after OTC. | At ovarian cryopreservation. Timeframe can be 1 to 15 years, an average of 3 years.
  Surgical bleedings above 500 mL in Turner syndrome females at cryopreservation
To examine occurrence of surgical complications after OTC. | At ovarian cryopreservation. Timeframe can be 1 to 15 years, an average of 3 years.
  The number of complications related to perforation of neighbouring organs.
To examine bone mineralization and body composition after OTC. | From the date of inclusion in study until autotransplantation. Timeframe can be up to 35 years.
  t-score at the DEXA scan
To examine quality of life (QoL) among participants. | At inclusion
  WHO QoL questionaire at inclusion (only girls > 15 years old)

CONTACTS AND LOCATIONS:
Locations (1):
- Mette Viuff, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No